CLINICAL TRIAL: NCT02474576
Title: Percutaneous Aponeurotomy in the Treatment of Dupuytren's Disease
Acronym: APADUP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Groupe Hospitalier Diaconesses Croix Saint-Simon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MMN_2015-1
Record Dates: First submitted 2015-06-12; First posted 2015-06-17 (Estimated); Last update posted 2021-02-11 (Actual); Status verified 2021-02

CONDITIONS: Dupuytren Disease
MeSH Terms: conditions — Dupuytren Contracture

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Percutaneous aponeurotomy (Experimental): Treatment of Dupuytrens-induced finger flessum using percutaneous aponeurotomy
  Interventions: Procedure: Percutaneous aponeurotomy

INTERVENTIONS:
Procedure: Percutaneous aponeurotomy — The finger(s) with limited extension due to Dupuytrens disease and for which the patient desires treatment, will be treated by fine-needle percutaneous aponeurotomy under local anesthesia (outpatient procedure). This procedure is already routinely used in clinical practice ; our study aims at better describing the time-sustainability of its benefits.

SUMMARY:
The efficiency of percutaneous aponeurotomy in the treatment of Dupuytrens disease is well known. However, the duration of the clinical improvement after aponeurotomy is not well known.

This study aims primarily at measuring the incidence rate of local relapse of Dupuytrens-induced finger flessum, within two years following treatment by percutaneous aponeurotomy in Dupuytrens.

ELIGIBILITY:
Inclusion Criteria:

* Patient suffers from Dupuytren disease
* Patient has at least one finger with at least 20° flessum on the metacarpophalangeal joint and/or on the proximal interphalangeal joint
* Patient has chosen to benefit from local treatment

Exclusion Criteria:

* Pregnancy
* Breastfeeding
* No social insurance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2019-04 (Actual); Study Completion 2020-04 (Actual)

PRIMARY OUTCOMES:
Frequency of local relapse at 24 months | 24 months after treatment by aponeurotomy
  the statistical unit is the finger treated by aponeurotomy (we expect an average of 2 fingers treated for one patient included). Local relapse is defined as the recurrence of a finger flessum superior by 20° to the articular range initially obtained after aponeurotomy

SECONDARY OUTCOMES:
Primary success rate of aponeurotomy | 3 months after treatment
  the statistical unit is the finger treated by aponeurotomy (we expect an average of 2 fingers treated for one patient included). Complete success is defined as a finger flessum inferior to 5°
Frequency of local relapse at 12 months | 12 months after treatment by aponeurotomy
Frequency of local relapse at 36 months | 36 months after treatment by aponeurotomy
Frequency of local relapse at 48 months | 48 months after treatment by aponeurotomy
Frequency of local relapse at 60 months | 60 months after treatment by aponeurotomy

CONTACTS AND LOCATIONS:
Locations (1):
- Diaconesses Croix Saint-Simon Hospital Group, Paris, France